CLINICAL TRIAL: NCT03546608
Title: Open-Label, Parallel-Group Phase 1 Study to Investigate the Effect of Various Degrees of Hepatic Impairment on the PK, Safety and Tolerability of the c-Met Kinase Inhibitor Tepotinib
Brief Title: Tepotinib Hepatic Impairment Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MS200095_0028
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-03

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; Tepotinib; Pharmacokinetics
MeSH Terms: interventions — tepotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Participants (Control) (Experimental): Participants with normal hepatic function matched to moderate hepatic impairment received single oral dose of 500 milligrams (mg) of tepotinib film-coated tablet on Day 1 after a standard breakfast.
  Interventions: Drug: Tepotinib
- Mild Hepatic Impairment (Child-Pugh Class A) (Experimental): Participants with mild hepatic impairment (Child-Pugh Class A, score 5 to 6) received single oral dose of 500 mg tepotinib film-coated tablet on Day 1 after a standard breakfast.
  Interventions: Drug: Tepotinib
- Moderate Hepatic Impairment (Child-Pugh Class B) (Experimental): Participants with moderate hepatic impairment (Child-Pugh Class B, score 7 to 9) received single oral dose of 500 mg tepotinib film-coated tablet on Day 1 after a standard breakfast.
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Participants received a single oral dose of tepotinib in Part 1.

SUMMARY:
The study investigated the effect of various degrees of hepatic impairment on the pharmacokinetics (PK), safety and tolerability of tepotinib.

ELIGIBILITY:
Inclusion Criteria:

* Men and women (of nonchildbearing potential), with a body mass index of 18 to 36 kilograms per meter square (inclusive) and a body weight greater than or equal to 50 kilograms at screening, with the absence of acute hepatitis or Human Immunodeficiency Virus 1 and 2, who gave informed consent and are willing and able to comply with study procedures were eligible for enrollment
* Participants with impaired hepatic function (Child-Pugh class A or Child-Pugh class B) and participants with normal hepatic function were eligible to enroll in the study
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Healthy participants were excluded if they have hepatitis B or C or had a previous infection with hepatitis C treated with Sofosbuvir or other antiviral compounds, or any other clinically relevant disease, as considered by the Investigator
* Participants with impaired hepatic function were excluded if they have primary biliary liver cirrhosis, nonstabilized chronic heart failure, hepatocarcinoma, hepatic encephalopathy (Grade III or IV), sepsis or gastrointestinal bleeding, or any other clinically relevant disease, as considered by the Investigator
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2019-02-05 (Actual); Study Completion 2019-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — EMD Serono Research & Development Institute, Inc., the biopharmaceutical division of Merck KGaA, Darmstadt, Germany
Locations (2):
- United States (2):
  - Qps Mra, Llc, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0028
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts: Part 1 and Part 2. Part 2 of the study was optional and sponsor decided not to perform part 2 of the study.
Period: Overall Study
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Started | 6 | 6 | 6
Completed | 6 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received tepotinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (8.0) | 61 (3.9) | 60 (10.0) | 60 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 4
  Male | 5 | 4 | 5 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 3 | 5 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 1 | 3
  White | 4 | 5 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity ( AUC0-inf ) of Tepotinib
Description: The area under the plasma concentration time curve (AUC) from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at the last sampling time (tlast), as estimated using the linear regression from lambda z determination. AUC(0- inf)=AUC0-t plus Clastpred/lambda z where Clastpred was last predicted concentration. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Pre-dose and 0.25, 0.5, 0.75, 1.0, 1.5, 2, 3, 4, 6, 8, 10, 12, 16, 24, 30, 36, 48, 54, 60, 72, 96, 120, 144, 168, 216, 288, 336 and 504 hours (for hepatic impaired participants only) post-dose on Day 1
Population: Pharmacokinetic (PK) Analysis Set included all participants who received a single dose of tepotinib and had at least 1 post-dose PK measurement without important protocol deviations/violations or events that could affect the PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram*hour per milliliter (ng*h/mL) | 27500 (13.4) | 26100 (63.9) | 24200 (26.9)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 94.99, 90% CI 2-sided [64.75 to 139.35]
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 87.92, 90% CI 2-sided [59.93 to 128.98]

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Tepotinib
Description: The AUC from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification (LLOQ). Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: as for outcome 1
Population: PK Analysis Set included all participants who received a single dose of tepotinib and had at least 1 post-dose PK measurement without important protocol deviations/violations or events that could affect the PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL | 27000 (13.8) | 25600 (65.6) | 23500 (27.4)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 94.81, 90% CI 2-sided [64.09 to 140.26]
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 87.20, 90% CI 2-sided [58.94 to 129.00]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib
Description: Maximum observed plasma concentration (Cmax) was taken directly from the observed concentration-time profile.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Nanogram per milliliter (ng/mL) | 406 (12.2) | 416 (31.5) | 288 (23.5)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 102.45, 90% CI 2-sided [80.90 to 129.73]
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 71.02, 90% CI 2-sided [56.08 to 89.93]

4. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Tepotinib
Description: Time to reach the maximum observed plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Hours | 11 [10.00 to 12.00] | 11.00 [8.00 to 24.00] | 16.00 [6.00 to 30.08]

5. Secondary Outcome: Apparent Terminal Half Life (t1/2) of Tepotinib
Description: Terminal half-life was calculated as log2 divided by lambda z. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Hours | 36.8 [32.3 to 48.4] | 43.7 [31.3 to 55.2] | 46.1 [41.9 to 74.4]

6. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Tepotinib
Description: Apparent total body clearance of drug from plasma following extravascular administration, calculated as dose/AUC0-infinity for tepotinib.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour | 16.4 (13.4) | 17.2 (63.9) | 18.6 (26.9)

7. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (VZ/f) of Tepotinib
Description: Apparent volume of distribution during the terminal phase following extravascular administration for tepotinib was calculated. Vz/f = Dose/(AUC0-infinity multiply by Lambda z) following single dose.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Liter | 892 (11.4) | 1050 (45.3) | 1400 (20.4)

8. Secondary Outcome: Extrapolated Area Under the Plasma Concentration-Time Curve From Time t to Infinity as a Percentage of AUC0-Inf (AUCextra) of Tepotinib
Description: AUCextra was defined as a percentage of AUC0-inf obtained by extrapolation: %AUCextra = (1- [AUC0-t/AUC0-inf])*100. %AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: as for outcome 1
Population: PK analysis set was used. Summary statistics for this parameter was not reported because it is a diagnostic parameter, rather than a PK parameter in the proper sense. It was only used to assess the individual data, not the group level. Therefore, individual data was reported for this outcome measure. Here, "Number Analyzed"= specific participant evaluated in respective arm.
Measure: Number; unit: Percentage of AUC0-inf
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of AUC0-inf
  Participant 1: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 | 1.34 | 5.01 | 3.35
  Participant 2: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 | 1.06 | 0.895 | 3.03
  Participant 3: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 | 2.14 | 1.33 | 1.49
  Participant 4: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 | 1.22 | 1.16 | 1.80
  Participant 5: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 | 2.45 | 1.55 | 1.60
  Participant 6: number analyzed (Participants) | 1 | 1 | 1
  Participant 6 | 2.08 | 1.41 | 3.87

9. Secondary Outcome: Extrapolated Area Under the Plasma Concentration-Time Curve From Time t to Infinity as a Percentage of AUC0-Inf (AUCextra) of Tepotinib Metabolite (MSC2571109)
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Number; unit: Percentage of AUC0-inf
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of AUC0-inf
  Participant 1: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 | 0.799 | 1.44 | 2.05
  Participant 2: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 | 1.28 | 0.574 | 1.41
  Participant 3: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 | 0.737 | 0.605 | 1.06
  Participant 4: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 | 0.677 | 0.470 | 3.06
  Participant 5: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 | 1.55 | 0.482 | 0.522
  Participant 6: number analyzed (Participants) | 1 | 1 | 1
  Participant 6 | 1.07 | 0.621 | 1.96

10. Secondary Outcome: Extrapolated Area Under the Plasma Concentration-Time Curve From Time t to Infinity as a Percentage of AUC0-Inf (AUCextra) of Tepotinib Metabolite (MSC2571107)
Description: as for outcome 8
Time Frame: as for outcome 1
Population: as for outcome 8
Measure: Number; unit: Percentage of AUC0-inf
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Percentage of AUC0-inf
  Participant 1: number analyzed (Participants) | 1 | 1 | 1
  Participant 1 | 0.592 | 3.69 | 2.10
  Participant 2: number analyzed (Participants) | 1 | 1 | 1
  Participant 2 | 0.925 | 0.848 | 5.68
  Participant 3: number analyzed (Participants) | 1 | 1 | 1
  Participant 3 | 0.671 | 0.516 | 0.683
  Participant 4: number analyzed (Participants) | 1 | 1 | 1
  Participant 4 | 0.639 | 0.513 | 3.08
  Participant 5: number analyzed (Participants) | 1 | 1 | 1
  Participant 5 | 1.77 | 0.731 | 2.45
  Participant 6: number analyzed (Participants) | 1 | 1 | 1
  Participant 6 | 0.904 | 1.15 | 1.97

11. Secondary Outcome: Area Under the Plasma Concentration Time Curve for Unbound Drug From Time Zero (Dosing Time) Extrapolated to Infinity (AUC0-inf, u) of Tepotinib
Description: Area under the concentration-time curve for unbound drug from time zero to infinity, calculated as AUC0-inf_pred multiplied by fu. Fu is the fraction of analyte unbound. Free fraction was calculated as the ratio of free concentration divided by total concentration at a given sampling point.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL | 532 (26.4) | 585 (40.5) | 653 (33.3)

12. Secondary Outcome: Maximum Observed Unbound Plasma Concentration (Cmax,u) of Tepotinib
Description: Maximum unbound plasma drug concentration, was calculated as Cmax*fu. Fu is the fraction of analyte unbound. Free fraction was calculated as the ratio of free concentration divided by total concentration at a given sampling point.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng/mL | 7.87 (25.6) | 9.32 (22.5) | 7.80 (22.3)

13. Secondary Outcome: Apparent Total Body Clearance of Unbound Drug Following Extravascular Administration (CL/f,u) of Tepotinib
Description: Unbound apparent oral clearance, was calculated as CL/f,u = Dose divided by AUC0-inf_pred/fu. Fu is the fraction of analyte unbound. Free fraction was calculated as the ratio of free concentration divided by total concentration at a given sampling point.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Liter per hour | 845 (26.4) | 770 (40.5) | 689 (33.3)

14. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-t) of Tepotinib Metabolites (MSC2571109 and MSC2571107)
Description: AUC0-t at which the concentration was at or above lower limit of quantification (LLOQ) was calculated according to the mixed log linear trapezoidal rule. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL
  MSC2571109 | 13300 (29.5) | 11000 (74.8) | 18100 (80.7)
  MSC2571107 | 1120 (34.1) | 1120 (88.8) | 1050 (70.4)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 82.62, 90% CI 2-sided [45.67 to 149.47] — For MSC2571109
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 136.59, 90% CI 2-sided [75.50 to 247.12] — For MSC2571109
Statistical Analysis 3: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 100.47, 90% CI 2-sided [54.53 to 185.10] — For MSC2571107
Statistical Analysis 4: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 94.48, 90% CI 2-sided [51.28 to 174.07] — For MSC2571107

15. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib Metabolites (MSC2571109 and MSC2571107)
Description: The area under the concentration time curve (AUC) from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at the last sampling time (tlast), as estimated using the linear regression from lambda z determination. AUC0-inf = AUC0-t plus Clastpred/lambda z where Clastpred was last predicted concentration. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng*h/mL
  MSC2571109 | 13400 (29.3) | 11100 (74.3) | 18500 (80.9)
  MSC2571107 | 1130 (33.7) | 1140 (87.2) | 1080 (69.2)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 82.35, 90% CI 2-sided [45.56 to 148.84] — For MSC2571109
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 137.51, 90% CI 2-sided [76.08 to 248.54] — For MSC2571109
Statistical Analysis 3: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 100.81, 90% CI 2-sided [55.16 to 184.23] — For MSC2571107
Statistical Analysis 4: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 96.18, 90% CI 2-sided [52.63 to 175.78] — For MSC2571107

16. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Tepotinib Metabolites (MSC2571109 and MSC2571107)
Description: Cmax was taken directly from the observed concentration-time profile.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
ng/mL
  MSC2571109 | 143 (33.9) | 132 (47.3) | 165 (37.9)
  MSC2571107 | 13.9 (39.2) | 14.8 (55.2) | 10.1 (32.1)
Statistical Analysis 1: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 92.30, 90% CI 2-sided [62.52 to 136.26] — For MSC2571109
Statistical Analysis 2: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 114.80, 90% CI 2-sided [77.76 to 169.48] — For MSC2571109
Statistical Analysis 3: Comparison: Healthy Participants (Control) vs Mild Hepatic Impairment (Child-Pugh Class A); Test type: Other; Ratio of Geometric Least Square Mean (%) = 106.51, 90% CI 2-sided [70.25 to 161.49] — For MSC2571107
Statistical Analysis 4: Comparison: Healthy Participants (Control) vs Moderate Hepatic Impairment (Child-Pugh Class B); Test type: Other; Ratio of Geometric Least Square Mean (%) = 72.58, 90% CI 2-sided [47.87 to 110.04] — For MSC2571107

17. Secondary Outcome: Time to Reach Maximum Observation Plasma Concentration (Tmax) of Tepotinib Metabolites (MSC2571109 and MSC2571107)
Description: as for outcome 4
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  MSC2571109 | 24.00 [24.00 to 48.00] | 24.00 [24.00 to 48.00] | 54.00 [24.00 to 72.00]
  MSC2571107 | 24.00 [24.00 to 30.00] | 24.00 [24.00 to 24.00] | 30.00 [16.00 to 72.00]

18. Secondary Outcome: Apparent Terminal Half Life (t1/2) of Tepotinib Metabolites (MSC2571109 and MSC2571107)
Description: as for outcome 5
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: Hours
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Hours
  MSC2571109 | 46.3 [43.9 to 56.4] | 57.5 [32.9 to 67.5] | 78.8 [55.5 to 128]
  MSC2571107 | 46.8 [43.8 to 58.6] | 40.7 [33.9 to 69.8] | 75.4 [53.3 to 137]

19. Secondary Outcome: Metabolite (MSC2571109 or MSC2571107) Area Under Curve From Time Zero Extrapolated To Infinity (AUC0-inf) to Tepotinib (AUC0-inf) Ratio
Description: The area under the concentration time curve (AUC) from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at the last sampling time (tlast), as estimated using the linear regression from lambda z determination. AUC0-inf = AUC0-t plus Clastpred/lambda z where Clastpred was last predicted concentration. Lambda z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve. Ratio of AUC0-inf of Metabolite (MSC2571109 or MSC2571107) to AUC0-inf of tepotinib was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Ratio
  MSC2571109 | 0.489 (31.8) | 0.424 (24.7) | 0.764 (49.5)
  MSC2571107 | 0.0410 (34.7) | 0.0435 (32.3) | 0.0449 (40.0)

20. Secondary Outcome: Metabolite (MSC2571109 or MSC2571107) Maximum Observed Plasma Concentration Observed (Cmax) to Tepotinib Cmax Ratio
Description: Cmax was taken directly from the observed concentration-time profile. Ratio of Cmax of Metabolite (MSC2571109 or MSC2571107) to Cmax of tepotinib was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Ratio
  MSC2571109 | 0.353 (27.5) | 0.318 (30.0) | 0.571 (37.3)
  MSC2571107 | 0.0343 (29.2) | 0.0357 (32.9) | 0.0351 (27.1)

21. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs included both serious TEAEs and non-serious TEAEs. Number of Participants with TEAEs were reported.
Time Frame: For Healthy Participants: Day 1 up to Day 15; For Hepatic Impaired Participants: Day 1 up to Day 22
Population: Safety Analysis Set included all participants who received tepotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 1 | 0 | 2

22. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameters
Description: Laboratory assessments included hematology, biochemistry, coagulation and urinalysis. Number of participants with clinically significant changes from baseline in laboratory parameters were reported. Clinical Significance was decided by the investigator.
Time Frame: For Healthy Participants: Day 1 up to Day 15; For Hepatic Impaired Participants: Day 1 up to Day 22
Population: Safety Analysis Set included all participants who received tepotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs and 12-lead Electrocardiogram (ECG) Findings
Description: Vital signs included body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. The 12-lead ECGs were recorded after the participants have rested for at least 5 minutes in supine position. Number of participants with clinically significant changes from baseline in vital signs and ECG were reported. Clinical Significance was decided by the investigator.
Time Frame: For Healthy Participants: Day 1 up to Day 15; For Hepatic Impaired Participants: Day 1 up to Day 22
Population: Safety Analysis Set included all participants who received tepotinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
Number analyzed (Participants) | 6 | 6 | 6
Participants
  Vital Signs | 0 | 0 | 0
  ECG Findings | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For Healthy Participants: Day 1 up to Day 15; For Hepatic Impaired Participants: Day 1 up to Day 22
Arm/Group | Healthy Participants (Control) | Mild Hepatic Impairment (Child-Pugh Class A) | Moderate Hepatic Impairment (Child-Pugh Class B)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Healthy Participants (Control) (N=6) | Mild Hepatic Impairment (Child-Pugh Class A) (N=6) | Moderate Hepatic Impairment (Child-Pugh Class B) (N=6)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT03546608/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/08/NCT03546608/SAP_001.pdf